CLINICAL TRIAL: NCT02543268
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Immunogenicity, Safety and Tolerability of a Heterologous Prime-Boost Regimen Using Three Different Batches of Ad26.ZEBOV and a Single Batch of MVA-BN®-Filo in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Immunogenicity, Safety and Tolerability of Ad26.ZEBOV and MVA-BN-Filo in Healthy Adult Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR107786; VAC52150EBL3003 (Other: Crucell Holland BV)
Record Dates: First submitted 2015-09-04; First posted 2015-09-07 (Estimated); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Healthy
Keywords: Ebola viruses; Ebola virus disease (EVD); Filoviruses; Monovalent vaccine; Safety; Immunogenicity; Human adenovirus serotype 26 (Ad26) expressing the Ebola virus Mayinga variant glycoprotein (Ad26.ZEBOV); Modified Vaccinia Virus Ankara - Bavarian Nordic Filo-vector (MVA-BN Filo); Healthy participants
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (4):
- Group 1 (Experimental): Ad26.ZEBOV -Batch #1, single dose intramuscular (IM) injection on Day 1; MVA-BN-Filo, single dose IM injection on Day 57
  Interventions: Biological: Ad26.ZEBOV-Batch #1; Biological: MVA-BN-Filo
- Group 2 (Experimental): Ad26.ZEBOV -Batch #2, single dose intramuscular (IM) injection on Day 1; MVA-BN-Filo, single dose IM injection on Day 57
  Interventions: Biological: Ad26.ZEBOV-Batch #2; Biological: MVA-BN-Filo
- Group 3 (Experimental): Ad26.ZEBOV -Batch #3, single dose intramuscular (IM) injection on Day 1; MVA-BN-Filo, single dose IM injection on Day 57
  Interventions: Biological: Ad26.ZEBOV-Batch #3; Biological: MVA-BN-Filo
- Group 4 (Experimental): Placebo (0.9% saline)- single dose IM injection on Day 1 and Day 57
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Ad26.ZEBOV-Batch #1 — Ad26.ZEBOV - Batch #1, live, replication incompetent vaccine, sterile suspension of 0.5 milliliter (mL) intramuscular (IM) injection of 5*10^10 viral particles on Day 1
  Arms: Group 1
Biological: Ad26.ZEBOV-Batch #2 — Ad26.ZEBOV - Batch #2, live, replication incompetent vaccine, sterile suspension of 0.5 milliliter (mL) intramuscular (IM) injection of 5*10^10 viral particles on Day 1
  Arms: Group 2
Biological: Ad26.ZEBOV-Batch #3 — Ad26.ZEBOV - Batch #3, live, replication incompetent vaccine, sterile suspension of 0.5 milliliter (mL) intramuscular (IM) injection of 5*10^10 viral particles on Day 1
  Arms: Group 3
Biological: MVA-BN-Filo — MVA-BN-Filo- live replication incompetent vaccine, 0.5 mL IM injection of 1*10^8 Infectious Unit [Inf. U.] once on Day 57.
  Arms: Group 1; Group 2; Group 3
Biological: Placebo — One 0.5 ml IM injection of 0.9% saline once on Day 1 and Day 57.
  Arms: Group 4

SUMMARY:
The purpose of this study is to compare the humoral immune response induced by 3 different batches of Ad26.ZEBOV as measured by enzyme - linked immunosorbent assay (ELISA) against the Ebola virus (EBOV) GP (Glycoprotein) at 56 days post prime.

DETAILED DESCRIPTION:
This is a randomized, double - blind, placebo - controlled, parallel - group, multicenter, Phase 3 study to evaluate the immunogenic equivalence of a heterologous prime - boost regimen using 3 different batches of Ad26.ZEBOV in healthy adult participants. The study consists of a screening period of up to 6 weeks, a vaccination period in which participants will be vaccinated at baseline (Day 1), followed by a boost vaccination on Day 57, and a post-vaccination phase until 6 months post-boost visit (Day 237). The participants will be randomized at baseline (on Day 1) in a 2:2:2:1 ratio to Groups 1, 2, 3 and 4. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy in the Investigator's clinical judgment on the basis of medical history, physical examination, electrocardiogram (ECG) and vital signs performed at Screening
* Healthy on the basis of clinical laboratory tests performed at Screening
* Before randomization, a woman must be either of childbearing potential and practicing (or intending to practice) a highly effective method of birth control consistent with local regulations regarding the use of birth control methods for participants participating in clinical studies, beginning at least 28 days prior to vaccination OR not of childbearing potential: postmenopausal (greater than [>] 45 years of age with amenorrhea for at least 2 years or any age with amenorrhea for at least 6 months, and a serum follicle stimulating hormone (FSH) level >40 international unit per milliliter [IU/L]); permanently sterilized (for example, bilateral tubal occlusion [which includes tubal ligation procedures as consistent with local regulations], hysterectomy, bilateral salpingectomy, bilateral oophorectomy); or otherwise be incapable of pregnancy
* Woman of childbearing potential must have a negative serum [beta-human chorionic gonadotropin (beta-hCG)] at Screening and a negative urine beta-hCG pregnancy test immediately prior to each study vaccine administration
* Man who is sexually active with a woman of childbearing potential and has not had a vasectomy performed more than 1 year prior to Screening must be willing to use condoms for sexual intercourse beginning prior to enrollment, in addition to the documented birth control method used by the female partner

Exclusion Criteria:

* Having received a candidate Ebola vaccine
* Diagnosed with Ebola virus disease, or prior exposure to Ebola virus, including travel to West Africa less than 1 month prior to Screening. West Africa includes but is not limited to the countries of Guinea, Liberia, Mali, and Sierra Leone
* Having received any experimental candidate adenovirus serotype 26 (vector: Ad26) or Modified Vaccinia Ankara (MVA-) based vaccine in the past
* Known allergy or history of anaphylaxis or other serious adverse reactions to vaccines or vaccine products (including any of the constituents of the study vaccines) including known allergy to egg, egg products and aminoglycosides
* Presence of acute illness or temperature greater than or equal to (>=) 38.0 centigrade (°C) on Day 1

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 329 (Actual)
Dates: Start 2015-09-21 (Actual); Primary Completion 2016-01-22 (Actual); Study Completion 2016-07-20 (Actual)

PRIMARY OUTCOMES:
Immune Responses to the Study Vaccine Regimens against Ebola virus (EBOV) Glycoprotein (GP) using EBOV GP protein enzyme-linked immunosorbent assay (ELISA) | At 56 days post prime vaccination
  The humoral immune response will be assessed by enzyme-linked immunosorbent assay (ELISA) binding antibody

SECONDARY OUTCOMES:
Immune Responses to the Study Vaccine Regimens against Ebola virus (EBOV) Glycoprotein (GP) using EBOV GP protein enzyme-linked immunosorbent assay (ELISA) | At Days 1, 29 post prime dose and at days 21, 42, and 180 post boost vaccination
  The humoral immune response will be assessed by enzyme-linked immunosorbent assay (ELISA) binding antibody
Number of Participants with Solicited Local and Systemic Adverse Events (AEs) | Up to 7 days after each vaccination
Number of Participants with Adverse Events (AEs) | Up to 42 days post boost vaccination
Number of Participants with Serious Adverse Events (SAEs) | Continuous throughout the duration of study (Up to 180 Days post boost vaccination)

CONTACTS AND LOCATIONS:
Overall Officials: Crucell Holland BV Clinical Trial, Study Director — Crucell Holland BV
Locations (6):
- United States (6):
  - Huntsville, Alabama
  - San Diego, California
  - Melbourne, Florida
  - Peoria, Illinois
  - Mishawaka, Indiana
  - Rockville, Maryland

REFERENCES:
- [Derived] Bockstal V, Gaddah A, Goldstein N, Shukarev G, Bart S, Luhn K, Robinson C, Anumendem D, Leyssen M, Douoguih M. Assessments of different batches and dose levels of a two-dose Ad26.ZEBOV and MVA-BN-Filo vaccine regimen. NPJ Vaccines. 2021 Dec 20;6(1):157. doi: 10.1038/s41541-021-00402-8. PMID 34930928